CLINICAL TRIAL: NCT06314295
Title: Automated Echocardiographic Detection of Coronary Artery Disease Using Artificial Intelligence Methods
Status: Recruiting | Type: Observational
Sponsor: Beijing Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: BeijingH-WF
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The incidence rate and mortality of coronary artery disease are increasing year by year. Exploring non-invasive, accurate, and widely applicable methods to screen and diagnosis is of great significance. New ultrasound techniques, such as non-invasive myocardial work, have been proven to be superior to traditional ultrasound techniques in screening and diagnosis. However, diagnostic analysis based on ultrasound video images is time-consuming and subjective. The progress of artificial intelligence technology in fully automated quantitative evaluation of video images provides the possibility for computer-aided design screening and diagnosis. At present, the application of artificial intelligence in computer-aided design is a cutting-edge issue in the field of cardiovascular disease research. The application of artificial intelligence technology in the construction of computer-aided diagnostic models based on ultrasound video images is still in its early stages.

DETAILED DESCRIPTION:
1) Clarify the value of new cardiac ultrasound techniques indicators in coronary artery disease diagnosis; 2) To achieve classification and detection of cardiac ultrasound sections; Implementing automatic segmentation and recognition of the left ventricular cavity, left ventricular myocardium, and left atrial wall contours through the CLAS model; Using the another model to achieve heart motion tracking and synthesizing velocity vector maps of the heart flow field. 3) Verify and optimize the coronary artery disease fully automated artificial intelligence diagnostic model mentioned above.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected coronary artery disease
* Patients plan to undergo coronary angiography

Exclusion Criteria:

* Patients with aortic valve stenosis
* Patients with aortic valve replacement surgery
* Patients with hypertrophic cardiomyopathy
* Patients with severe heart valve disease
* Patients with severe arrhythmia
* Patients with severe cardiomyopathy
* Patients with severe congenital heart disease
* The quality of ultrasound images is poor

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with suspected coronary artery disease who plan to undergo coronary angiography
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2026-03-11 (Estimated); Study Completion 2026-05-11 (Estimated)

PRIMARY OUTCOMES:
Different coronary angiography results | Coronary angiography examination within 2-3 days after admission
  The degree of coronary artery stenosis

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Hospital, Beijing, China